CLINICAL TRIAL: NCT05153707
Title: Evaluation of a Clinical Pharmacist-led Discharge Education Service in Patients With Acute Coronary Syndrome: A Randomized Controlled Study
Brief Title: Clinical Pharmacist-led Discharge Education Service in Acute Coronary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Betul Okuyan, Assoc.Prof., Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MARCPD-0001
Record Dates: First submitted 2021-11-25; First posted 2021-12-10 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical Pharmacist-led discharge education program (Experimental): Clinical pharmacist-led services
  Interventions: Behavioral: Discharge Education Program
- Control group (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Discharge Education Program — medication reconciliation, medication review, individually prepared patient medicine (pill) card, patient education (based on Health Belief Model by using written material and video, and verbally [by using Teach back method especially for patients with low health literacy]) and counseling (using behavior change techniques based on The Capability, Opportunity, and Motivation Behavior model).
  Arms: Clinical Pharmacist-led discharge education program

SUMMARY:
To evaluate the impact of clinical pharmacist-led discharge education service in patients with acute coronary syndrome.

DETAILED DESCRIPTION:
This prospective, randomized controlled study was conducted in patients with acute coronary syndrome in an cardiology service of tertiary training and research hospital. The clinical pharmacist, within the scope of the discharge education services, provided medication reconciliation, medication review, individually prepared patient medicine (pill) card, patient education (based on Health Belief Model by using written material and video, and verbally [by using Teach back method especially for patients with low health literacy]) and counseling (using behavior change techniques based on The Capability, Opportunity, and Motivation Behavior model). The control group received standard care.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the cardiology department due to acute coronary syndrome
* Older than 18 years old

Exclusion Criteria:

* Patients who transferred to another ward
* Patients with active malignancy
* Patients with alzheimer and/or dementia diagnosis
* Patient with >%80 visual loss or deaf muteness reported at medical record

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
30 days hospital re-admission for cardiac reasons | 30 days
  Proportion of patients readmitted to hospital for cardiac cause at 1 month

SECONDARY OUTCOMES:
Hospital re-admission for cardiac reasons | 3 months, 6 months, and 12 months
  Proportion of patients readmitted to hospital for cardiac cause through 1 year.
Hospital re-admission for any reasons | 1 month, 3 months, 6 months, and 12 months
  Proportion of patients readmitted to hospital for any cause through 1 year.
Emergency service visits | 1 month, 3 months, 6 months, and 12 months
  Proportion of patients visited to emergency service through 1 year.
Major Adverse Cardiovascular Event | 1 month, 3 months, 6 months, and 12 months
  Proportion of patients had major adverse cardiovascular event through 1 year.
Death for cardiac reason | 1 month, 3 months, 6 months, and 12 months
  Proportion of patients died for cardiac cause through 1 year.
Death for any reason | 1 month, 3 months, 6 months, and 12 months
  Proportion of patients dying for any cause through 1 year.
Medication Adherence | 1 month, 3 months, 6 months, and 12 months
  Adherence to Cardioprotective Medications (Clopidogrel, Statins, Beta-blockers, Angiotensin-converting enzyme (ACE) inhibitors/ Angiotensin receptor blocker (ARB) through 1 year assessed by Medication Adherence Report Scale (MARS). MARS assesses adherence through 5-item, summed to give a scale score ranging from 5 to 25, where higher scores indicate higher levels of reported adherence.
Quality of Life Measurement | 1 month, 3 months, 6 months, and 12 months
  Change in quality of life from baseline assessed with EuroQol questionnaire EQ-5D-3L through 1 year. (EQ-5D-3L) is a standardized scale for use as a measure of the quality of life. The EQ-5D-3L descriptive system comprises the following 5 dimensions (5D): mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 3 levels (3L): no problems (1 point), some problems (2 points), extreme problems (3 points).
  This gives a total of 245 different health states, adding unconscious and dead.
Achieved Target Low-density Lipoprotein Value | 6 months, 12 months
  Rate of patients achieved target low-density lipoprotein value

CONTACTS AND LOCATIONS:
Overall Officials: Betul Okuyan, Principal Investigator — Marmara University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No